CLINICAL TRIAL: NCT00097526
Title: Bone Mineral Density in Adolescent Subjects With Growth Hormone Deficiency Who Are Completing Treatment With Nutropin AQ, Nutropin, or Protropin in the National Cooperative Growth Study (NCGS)
Brief Title: Bone Mineral Density (BMD) in Adolescents With Growth Hormone Deficiency (GHD)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 85-036, Substudy 10
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Dwarfism, Pituitary; Turner Syndrome
Keywords: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, open-label, postmarketing surveillance study. The substudy will collect information on BMD in adolescents and young adults with GHD or Turner syndrome who are completing GH treatment for statural indications.

ELIGIBILITY:
Inclusion Criteria:

* Bone age of at least 15 years for girls or at least 16 years for boys within 6 months of obtaining the DXA scan
* Previous enrollment in the NCGS core study, 85-036
* Tanner Stage 4 or greater
* Either spontaneous or induced puberty
* Subjects who plan on terminating GH treatment for statural purposes for one or more of the following reasons: epiphyseal fusion, slowing growth rate indicates that near adult height has been reached, or satisfied with current height

Exclusion Criteria:

* Current therapy with a non Genentech GH product
* Pregnancy (to avoid exposure to low levels of radiation from DXA scanners)
* Bilateral hip replacement
* Weight >130 kg (286 lb.)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2000-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lippe, M.D., Study Director — Genentech, Inc.